CLINICAL TRIAL: NCT02286206
Title: A Pilot Study to Determine How Frequency of Administration Modifies Steady-State Plasma Concentrations of Orally Administered Clozapine
Brief Title: Study of the Effect of Dosing on Clozapine Levels
Acronym: PK-CLZ
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ric Procyshyn, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H14-01644
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: Clozapine; Psychotropic Drugs; Antipsychotic Agents; Psychotic Disorders; Schizophrenia; Adverse Effects; Drug Monitoring
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clozapine bid (Experimental): Participants have been taking clozapine once daily and have reached steady-state prior to the start of this study.
  Intervention: Days 1-14
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine — One-half baseline dose po bid (or one-third baseline dose po qam and two-thirds baseline dose po qhs at the discretion of the treating clinicians and principal investigator)
  Other Names: Clozaril; FazaClo

SUMMARY:
The objectives of this 15-day study are:

1. To compare steady-state trough plasma concentrations of clozapine and its metabolite norclozapine when given once daily and twice daily (at the same total daily dose)
2. To determine if frequency of clozapine administration has an effect on:

   1. Symptoms of schizophrenia
   2. Adverse effects of clozapine
   3. Fasting blood glucose, lipids, creatinine, and urea
   4. Weight and waist circumference

DETAILED DESCRIPTION:
It is important that clinicians do everything possible to optimize the use of clozapine in individuals with treatment-resistant schizophrenia. To our knowledge, there are no published studies evaluating whether twice daily administration of clozapine is better than once daily administration in terms of effectiveness and tolerability. Although this may seem trivial at first, when we consider that clozapine has a relatively short half-life and dissociates quickly from the dopamine D2 receptor, it justifies further consideration. It takes on even more significance knowing that the established threshold clozapine plasma concentration for therapeutic response (i.e., 350-420 ng/ml) was determined using steady-state trough plasma samples (i.e., approximately 12 hours after the evening dose) in patients administered clozapine twice rather than once daily.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 19 - 65
* Participants must be fluent in English
* Participants must have a psychiatric diagnosis and are currently treated with clozapine once daily in the evening
* Participants must be on a stable dose of clozapine for at least one week to ensure steady-state has been achieved

Exclusion Criteria:

* Participants who are hypersensitive to clozapine
* Participants who are pregnant or lactating
* Participants who are of childbearing age and not using reliable contraception
* Participants who have postsurgical complications of the gastrointestinal tract that might impair absorption
* Participants who have any clinically relevant abnormalities of laboratory parameters
* Participants who have had a potent CYP1A2 metabolic inducer (e.g., carbamazepine; rifampin) or inhibitor (e.g., amiodarone; cimetidine; efavirenz; fluoroquinolone antibiotics; ticlopidine) added to and/or removed from their medication regimen in the past two weeks

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in steady-state trough plasma concentrations of clozapine and norclozapine at Days 7 and 14. | Days 0 (baseline), 7, and 14
  Steady-state trough plasma concentrations of clozapine and norclozapine will be measured on Days 7 and 14 and compared to those obtained on Day 0 (baseline).

SECONDARY OUTCOMES:
Change from baseline in symptoms at Day 14. | Day 0 (baseline) and 14
  As assessed by structured clinical interviews for the Positive and Negative Syndrome Scale (PANSS)
Change from baseline in side effect burden at Day 14 | Days 0 (baseline) and 14
  As assessed by the Udvalg for Kliniske Undersøgelser (UKU) Side Effect Rating Scale
Changes from baseline in laboratory measures at Day 14. | Days 0 (baseline) and 14
  Laboratory measures include fasting blood glucose, fasting lipid profile, creatinine, and urea.
Change from baseline in weight and waist circumference at Day 14. | Days 0 (baseline) and 14

CONTACTS AND LOCATIONS:
Overall Officials: Ric M. Procyshyn, Ph.D, Principal Investigator — University of British Columbia; Alasdair Barr, Ph.D, Study Director — University of British Columbia; William Honer, MD, Study Director — University of British Columbia; Randall White, MD, Study Director — University of British Columbia
Locations (1):
- UBC Hospital - Detwiller Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No